CLINICAL TRIAL: NCT03172793
Title: Pharmacokinetics and Tolerability of Telavancin at Differing Dosing Regimens in Cystic Fibrosis Adults Admitted With Acute Pulmonary Exacerbations
Brief Title: Telavancin Pharmacokinetics in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph L. Kuti, PharmD (Other)
Collaborators: Cumberland Pharmaceuticals, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Joseph L. Kuti, PharmD, Associate Director, CAIRD, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HHC-2017-0093
Record Dates: First submitted 2017-05-09; First posted 2017-06-01 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Cystic Fibrosis
Keywords: telavancin; lipoglycopeptide; MRSA; pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis | interventions — telavancin

STUDY DESIGN:
Intervention Model Description: This pharmacokinetic study uses a sequential, adaptive design to determine the pharmacokinetics and safety/tolerability of increasing weight based doses of telavancin. During Arm 1, participants will receive 7.5 mg/kg daily. Upon completion of data collection and assessment of safety/tolerability, Arm 2 participants will receiving 10 mg/kg daily. After completion of Arms 1 and 2, a preliminary pharmacokinetic and pharmacodynamic analysis will be conducted. These results, combined with the safety/tolerability of the 10mg/kg dose, will provide decision support to select a PK/PD optimized dose for Arm 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Telavancin injection Dose 1 (7.5mg/kg) (Experimental): The pharmacokinetics and tolerability of telavancin 7.5mg/kg q24h will be measured in 6 participants.
  Interventions: Drug: Telavancin Injection
- Telavancin injection Dose 2 (10mg/kg) (Experimental): After completion and analysis of 7.5mg/kg group, the next 6 participants will receive 10mg/kg q24h, and pharmacokinetics and tolerability will be measured.
  Interventions: Drug: Telavancin Injection
- Telavancin injection Dose 3 (TBD) (Experimental): The third arm will enroll 6 participants to receive the following dose of telavancin q24h: 7.5, 10, 12.5, or 15 mg/kg. The final dose will be selected based on pharmacokinetic studies from first 12 participants, tolerability, and pharmacodynamic modeling.
  Interventions: Drug: Telavancin Injection

INTERVENTIONS:
Drug: Telavancin Injection — Receive 3 doses of telavancin as described in arm/groups, followed by collection of blood for pharmacokinetic analyses.
  Other Names: Vibativ

SUMMARY:
Due to emerging resistance, new antibiotic options are needed to treat CF acute pulmonary exacerbations caused by methicillin resistant Staphylococcus aureus (MRSA). There is established evidence that adult patients with cystic fibrosis (CF) may have altered antibiotic pharmacokinetics compared with non-CF patients. Telavancin is a lipoglycopeptide antibiotic that has activity against gram-positive bacteria including MRSA. This study will determine the pharmacokinetics and tolerability of telavancin in 18 adult CF patients admitted for a pulmonary exacerbation at 1 of 4 participating hospitals in the US.

DETAILED DESCRIPTION:
Each participant will receive 3 doses of intravenous telavancin administered every 24 hours. Up to three different doses of telavancin will be studied (n=6 per group). Blood samples will be collected throughout the study to determine the pharmacokinetics of telavancin. Each group will proceed after measurement of safety, tolerability, and pharmacokinetics of the lower dose group before it.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Documented diagnosis of CF
* Acute pulmonary exacerbation as the primary reason for admission to the hospital with requirement to receive systemic antibiotic treatment, as defined by treating provider
* If female, subjects must be non-pregnant and non-lactating. Females can be either not of a child-bearing potential or if of a child-bearing potential, on acceptable modes of birth control such as abstinence from sexual intercourse, oral/parenteral contraceptives, or barrier method

Exclusion Criteria:

* History of any moderate or severe hypersensitivity or allergic reaction to telavancin or any component of telavancin, or any glycopeptide (e.g., vancomycin) antibiotic (a history of red man syndrome with vancomycin is not an exclusion criteria)
* History of any solid organ transplantation within the last 12 months
* Moderate to severe renal dysfunction defined as a creatinine clearance (CLCR) < 50 mL/min (as calculated by the Cockcroft-Gault equation using actual body weight) or requirement for continuous renal replacement therapy or hemodialysis
* Oliguria (urine output < 0.4 mL/kg/hr for at least 12 hours, up to a total of <20 mL/hr) or significant alterations in fluid/electrolyte homeostasis in a 72 hour window before enrollment with a history of renal compromise
* A hemoglobin less than 8 gm/dl at baseline
* Anticipated length of hospital stay less than 4 days, which would prevent completion of dose administration and pharmacokinetic sampling
* Receiving intravenous vancomycin at the time of enrollment or anticipation of requiring intravenous vancomycin during study participation (Note. Other antibiotics targeting Gram-positive bacteria such as MRSA are permitted)
* Receiving an anticoagulant AND requires specific coagulation testing (prothrombin time/international normalized ratio, activated partial thromboplastin time, activated clotting time, or coagulation based factor x activity assay) within 24 hours of receiving a telavancin dose (Note. Although telavancin does not interfere with coagulation, it may interfere with some assays used to monitor coagulation)
* Requirement of concomitant administration of agents containing a cyclodextrin solubilizer such as intravenous voriconazole or itraconazole
* Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)
* Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data
* Planned or prior participation in any other interventional drug study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Telavancin Clearance | 1, 24, 25, 48, 49-49.08, 49.25-49.5, 50-51, 52-53, 55-56, 57-61, and 72 hours after start of dosing.
  This outcome measures the total body clearance (L/hr) of telavancin over the 4 day study.
Telavancin Volume of Distribution | 1, 24, 25, 48, 49-49.08, 49.25-49.5, 50-51, 52-53, 55-56, 57-61, and 72 hours after start of dosing.
  This outcome measures the volume of distribution (L) of telavancin over the 4 day study.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 4 days
  This outcome measures the safety and tolerability of telavancin over the 4 day study with specific attention to changes in chemistry, complete blood count, and liver function tests before and after treatment, as well as any participant reported adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Kuti, PharmD, Principal Investigator — Hartford Hospital
Locations (5):
- United States (5):
  - Hartford Hospital, Hartford, Connecticut
  - IU Health University Hospital, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - St. Christophers Hospital for Children, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Shadyside, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kidd JM, Sakon CM, Oleksiuk LM, Cies JJ, Pettit RS, Nicolau DP, Kuti JL. Pharmacokinetics of Telavancin in Adult Patients with Cystic Fibrosis during Acute Pulmonary Exacerbation. Antimicrob Agents Chemother. 2019 Dec 20;64(1):e01914-19. doi: 10.1128/AAC.01914-19. Print 2019 Dec 20. PMID 31685468